CLINICAL TRIAL: NCT03612258
Title: Brain Mechanisms of Altered Sensory Perception and Self-Referential Processing in Juvenile Fibromyalgia
Brief Title: Brain Mechanisms of Juvenile Fibromyalgia
Acronym: JFM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Principal Investigator, Robert Coghill, Professor, Children's Hospital Medical Center, Cincinnati
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CIN_brainjfm_001
Record Dates: First submitted 2018-07-26; First posted 2018-08-02 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2025-01

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; Pain; Neuroimaging; Sensory sensitivity; Fatigue
MeSH Terms: conditions — Fibromyalgia; Pain; Fatigue | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Functional Magnetic Resonance Imaging (Experimental)
  Interventions: Diagnostic Test: Functional Magnetic Resonance Imaging

INTERVENTIONS:
Diagnostic Test: Functional Magnetic Resonance Imaging — Functional Magnetic Resonance Imaging scans will be completed to assess neural responses to painful, non-painful sensory, and emotion-eliciting stimuli.

SUMMARY:
This study evaluates whether differences exist between adolescent females with juvenile-onset fibromyalgia and healthy controls in processing of pain and emotion at the neural level as assessed by functional magnetic resonance imaging (fMRI). The study includes a longitudinal component to evaluate changes in neural processing of pain and emotion before and after different treatment strategies.

DETAILED DESCRIPTION:
Juvenile-onset fibromyalgia (JFM) is a chronic, widespread pain condition that primarily affects females. Previous work has shown increased sensitivity to painful and non-painful sensory stimuli in adults with fibromyalgia, as well as brain processing abnormalities associated with these stimuli. These abnormalities in adults are highly predictive of fibromyalgia status (as opposed to healthy status) in adults. Although JFM has some similar symptoms and features to fibromyalgia in adults, the neural mechanisms of JFM may be partially different, given the moment of sharp brain development characterising JFM. fMRI scans will be completed before and after different treatments for JFM (e.g. neuromuscular training + cognitive behavioral therapy, graded aerobic exercise) to investigate the effects of treatment on brain measures related to pain, fatigue and emotion processing.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Juvenile Fibromyalgia (by a pediatric rheumatologist or pain physician using 2010 American College of Rheumatology criteria)
* Right handed
* Functional Disability Index score ≥ 7, indicating at least mild disability
* Stable medication regimen for 3 weeks prior to MRI scan

Exclusion Criteria:

* Non-MRI compatible metal objects in the body (including braces, permanent upper retainers)
* Comorbid rheumatic disease (e.g. juvenile arthritis, systemic lupus erythematosus)
* Major psychiatric diagnoses (e.g. bipolar disorder, obsessive compulsive disorder, schizophrenia) or documented developmental delay
* Taking opioid pain medication

Ages: 13 Years to 17 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 153 (Actual)
Dates: Start 2018-02-28 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Functional brain activation differences | Baseline
  Functional Magnetic Resonance Imaging: differences in pain processing and emotional processing relative to healthy controls

SECONDARY OUTCOMES:
Functional brain activation differences | Baseline and 8 weeks
  Functional Magnetic Resonance Imaging: differences in response to painful, non-painful sensory, and emotion-eliciting stimuli before and after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Robert Coghill, PhD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
We plan to share behavioral MRI task data and functional brain imaging data, after the main results of the study have been published.
Supporting Information: Study Protocol
Time Frame: Data will become available after main study results (data from primary outcomes/aims of the study) have been published

REFERENCES:
- [Derived] Tong H, Maloney TC, Payne MF, Sunol M, Dudley JA, King CD, Ting TV, Kashikar-Zuck S, Coghill RC, Lopez-Sola M. Augmented pain-evoked primary sensorimotor cortex activation in adolescent girls with juvenile fibromyalgia. Pain. 2023 Oct 1;164(10):2316-2326. doi: 10.1097/j.pain.0000000000002933. Epub 2023 Jun 16. PMID 37326678